CLINICAL TRIAL: NCT04953312
Title: Calprotectin Involvement in Emergency Hematopoiesis Observed in Severe COVID-19
Brief Title: Calprotectin, a Biomarker of COVID-19 Severity (CALPRO)
Acronym: CALPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210522; 2021-A00674-37 (Other: ID-RCB Number)
Record Dates: First submitted 2021-07-05; First posted 2021-07-07 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Severe/Moderate Coronavirus; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Old Age
Keywords: Calprotectin; hematopoiesis; COVID-19
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 patients (group 1) (Experimental): Patients with a recent diagnosis (<7 days since first symptoms) of moderate or severe COVID-19
  Interventions: Biological: Blood samples
- Chronic myeloid malignancies (group 2) (Experimental): Adults with chronic myeloid malignancies including myelodysplastic syndromes with low risk MDS ; high risk MDS according to IPSS-R or with dysplastic or proliferative chronic myelomonocytic leukemia according to WHO2016
  Interventions: Biological: Blood samples
- Control group (group 3) (Other): Age-matched healthy donors
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — blood

SUMMARY:
The purpose of this study is to provide new insights into the pathophysiology of emergency hematopoiesis detected in severe COVID-19 patients. The investigators aim to explore the ability of calprotectin to induce an immunosuppressive myeloid program at the hematopoietic stem and progenitor cell (HSPC) level, and to identify the receptor(s) involved in this effect. Since patients with a hematological malignancy demonstrate a very high propensity to develop a severe COVID-19, the investigators will explore how HSPCs collected from patients with a myeloid malignancy respond to calprotectin.

DETAILED DESCRIPTION:
Emergency myelopoiesis in response to SARS-CoV-2 infection produce immunosuppressive myeloid cells with accumulation of immature granulocytes and loss of non-classical monocytes. Excessive release of calprotectin, the dimer of S100A8/A9 alarmins, by immature granulocytes and activated monocytes reflects this situation. A role of calprotectin has been previously described in the initiation and progression of chronic hematological malignancies such as myelodysplastic syndromes.

To provide a rationale for the targeting of alarmin-driven signaling pathways and limit the pathogenic inflammatory response to SARS-CoV-2 infection, the role of calprotectin in the production of immunosuppressive cells from the bone marrow hematopoietic stem and progenitors cells needs to be investigated in patients with severe COVID-19 in comparison with patients with chronic myeloid malignancies (such as chronic myelomonocytic leukemia and myelodysplastic syndromes) and with age-mached healthy controls.

A comprehensive and integrated multiomics approach will be used to decipher the features of immunosuppressive cells and identify therapeutic targets in deregulated pathways.

ELIGIBILITY:
Inclusion Criteria:

Criteria for all groups:

* Adults ≥ 18 years
* Dated and signed inform consent *

  * * : written informed consent of relative (trusted person, close family) in case of emergency procedure, by default emergency inclusion notified in medical file and pursuance consent sought.
* Affiliation with a social security scheme

Criteria for control group:

* Age-matched healthy donors

Criteria for chronic myeloid malignancies:

* A diagnosis of low or high-risk myelodysplastic syndromes according to the WHO 2016 classification
* A diagnosis of dysplastic or proliferative chronic myelomonocytic leukemia according to WHO 2016

Criteria for COVID-19 patients:

* Patients with a recent diagnosis (<7 days since first symptoms) of moderate or severe COVID-19

Exclusion Criteria:

* Pregnant women
* Minor patient or major under protection
* Patients with COVID-19 infection and active cancer or a history of cancer within the last 6 months
* Patients with COVID-19 and severe comorbidities including cardiovascular or respiratory diseases, unbalanced diabetes, obesity (IMC >29)
* Patient on AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Differential gene expression and epigenetic signature of COVID-19 or leukemic versus normal HSC using CITE-seq and ATAC-seq | 12 months
  Hematopoietic stem and progenitor cells from patients with severe or moderate COVID-19 or chronic myeloid malignancies or controls will be purified for analyses of transcriptome and chromatin conformation, and also functionally characterized using in vitro culture systems. Results will be compared between the three groups.

SECONDARY OUTCOMES:
Ex vivo testing of calprotectin-receptor interaction inhibitor | During the last 6 months of the study
  Expression of targeted receptors will be monitored by flow cytometry. Clinically developed compounds that could inhibit calprotectin effects will be tested in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela FONTENAY, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Eric SOLARY, MD, Study Director — Gustave Roussy Institut
Locations (1):
- Gustave Roussy Institut, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silvin A, Chapuis N, Dunsmore G, Goubet AG, Dubuisson A, Derosa L, Almire C, Henon C, Kosmider O, Droin N, Rameau P, Catelain C, Alfaro A, Dussiau C, Friedrich C, Sourdeau E, Marin N, Szwebel TA, Cantin D, Mouthon L, Borderie D, Deloger M, Bredel D, Mouraud S, Drubay D, Andrieu M, Lhonneur AS, Saada V, Stoclin A, Willekens C, Pommeret F, Griscelli F, Ng LG, Zhang Z, Bost P, Amit I, Barlesi F, Marabelle A, Pene F, Gachot B, Andre F, Zitvogel L, Ginhoux F, Fontenay M, Solary E. Elevated Calprotectin and Abnormal Myeloid Cell Subsets Discriminate Severe from Mild COVID-19. Cell. 2020 Sep 17;182(6):1401-1418.e18. doi: 10.1016/j.cell.2020.08.002. Epub 2020 Aug 5. PMID 32810439
- [Background] Shi H, Zuo Y, Yalavarthi S, Gockman K, Zuo M, Madison JA, Blair C, Woodward W, Lezak SP, Lugogo NL, Woods RJ, Lood C, Knight JS, Kanthi Y. Neutrophil calprotectin identifies severe pulmonary disease in COVID-19. J Leukoc Biol. 2021 Jan;109(1):67-72. doi: 10.1002/JLB.3COVCRA0720-359R. Epub 2020 Sep 1. PMID 32869342
- [Background] Udeh R, Advani S, de Guadiana Romualdo LG, Dolja-Gore X. Calprotectin, an Emerging Biomarker of Interest in COVID-19: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Feb 15;10(4):775. doi: 10.3390/jcm10040775. PMID 33672040
- [Background] Abers MS, Delmonte OM, Ricotta EE, Fintzi J, Fink DL, de Jesus AAA, Zarember KA, Alehashemi S, Oikonomou V, Desai JV, Canna SW, Shakoory B, Dobbs K, Imberti L, Sottini A, Quiros-Roldan E, Castelli F, Rossi C, Brugnoni D, Biondi A, Bettini LR, D'Angio' M, Bonfanti P, Castagnoli R, Montagna D, Licari A, Marseglia GL, Gliniewicz EF, Shaw E, Kahle DE, Rastegar AT, Stack M, Myint-Hpu K, Levinson SL, DiNubile MJ, Chertow DW, Burbelo PD, Cohen JI, Calvo KR, Tsang JS; NIAID COVID-19 Consortium; Su HC, Gallin JI, Kuhns DB, Goldbach-Mansky R, Lionakis MS, Notarangelo LD. An immune-based biomarker signature is associated with mortality in COVID-19 patients. JCI Insight. 2021 Jan 11;6(1):e144455. doi: 10.1172/jci.insight.144455. PMID 33232303
- [Background] Bauer W, Diehl-Wiesenecker E, Ulke J, Galtung N, Havelka A, Hegel JK, Tauber R, Somasundaram R, Kappert K. Outcome prediction by serum calprotectin in patients with COVID-19 in the emergency department. J Infect. 2021 Apr;82(4):84-123. doi: 10.1016/j.jinf.2020.11.016. Epub 2020 Nov 17. No abstract available. PMID 33217473
- [Background] Luis Garcia de Guadiana Romualdo, Mulero MDR, Olivo MH, Rojas CR, Arenas VR, Morales MG, Abellan AB, Conesa-Zamora P, Garcia-Garcia J, Hernandez AC, Morell-Garcia D, Dolores Albaladejo-Oton M, Consuegra-Sanchez L. Circulating levels of GDF-15 and calprotectin for prediction of in-hospital mortality in COVID-19 patients: A case series. J Infect. 2021 Feb;82(2):e40-e42. doi: 10.1016/j.jinf.2020.08.010. Epub 2020 Aug 12. No abstract available. PMID 32795482
- [Background] Mahler M, Meroni PL, Infantino M, Buhler KA, Fritzler MJ. Circulating Calprotectin as a Biomarker of COVID-19 Severity. Expert Rev Clin Immunol. 2021 May;17(5):431-443. doi: 10.1080/1744666X.2021.1905526. Epub 2021 Apr 13. PMID 33750254
- [Background] Kaya T, Yaylaci S, Nalbant A, Yildirim I, Kocayigit H, Cokluk E, Sekeroglu MR, Koroglu M, Guclu E. Serum calprotectin as a novel biomarker for severity of COVID-19 disease. Ir J Med Sci. 2022 Feb;191(1):59-64. doi: 10.1007/s11845-021-02565-8. Epub 2021 Feb 27. PMID 33641087
- See also: Groupe Francophone des Myélodysplasies: GFM is a cooperative group of the French Society of Hematology — http://www.gfmgroup.org